CLINICAL TRIAL: NCT05241106
Title: a Single-arm, Open, Multicenter, Phase II Study to Investigator the Efficacy and Safety of HYML-122 in Patients With FLT3 Positive Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Study of HYML-122 in Patients With FLT3 Positive Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tarapeutics Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYML-122-02
Record Dates: First submitted 2022-01-16; First posted 2022-02-15 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HYML-122 treatment (Experimental): HYML-122 tablets, 200mg spec, 28 days for each cycle. The first eligible three enrolled subjects will be administrated with 600mg bid dose regimen for 28 consecutive days ( 1 treatment cycle). The Data Monitoring Committee (DMC) will evaluate the safety, efficacy and PK data of these three subjects and make decision whether the regimen need to be adjusted (increasing/decreasing administration dosing or adjusting dosing frequency).
  Interventions: Drug: HYML-122

INTERVENTIONS:
Drug: HYML-122 — each treatment cycle is comprised of 28-day consecutive dosing of HYML-122. Upon completion of each cycle, patients may continue to receive oral HYML-122 tablets if they are benefit from the treatment and the toxicity is tolerable.

SUMMARY:
this is a single-arm, open, multicenter, phase 2 study to evaluate the efficacy, safety and pharmacokinetics of HYLM-122 monotherapy in Chinese subjects with FLT3 positive relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the procedures of the clinical study and participate voluntarily with signed and dated written informed consent form, comply with the requirements of the study protocol.
* Males and/or females at least 18 years old when signing the informed consent form.
* Histologically confirmed AML (defined using WHO criteria 2016) with one of the following:

Refractory to at least 1 cycle of induction chemotherapy. Relapsed after achieving remission with a prior therapy.

* Subject is positive for FLT3 mutation in bone marrow or blood after completion of the subject's last interventional treatment.
* Eastern cooperative oncology group performance status (ECOG) ≤2 at screening.
* Life expectancy of at least 3 months.
* Women of childbearing potential have a negative pregnancy test at baseline and are willing to employ an effective method of contraception for the entire duration of study treatment and 6 months after the last dose.

Exclusion Criteria:

* Known or suspected allergies to any of the investigational drug composition (HYML-122, lactose, hydroxypropyl cellulose, hyposubstituted hydroxypropyl cellulose, silicon dioxide, magnesium stearate, titanium dioxide and polyethylene glycol).
* Medical history and surgical history excluded according to the protocol.
* Any previous medical treatment history exclude from the protocol.
* Abnormal laboratory results exclude from the protocol.
* Combination of treatments and/or drugs required during the study period and cannot be discontinued that excluded from the protocol.
* Alcohol abuse within 6 months prior to screening, defined as long-term drinking history, generally more than 5 years, equivalent to alcohol quantity ≥40g/d for men, ≥20g/d for women, or heavy drinking history within 2 weeks, equivalent to alcohol quantity ≥80g/d. alcohol volume (g) conversion formula=alcohol consumption (mL)*alcohol content (%)*0.8.
* Abortion less than 30 days prior to screening, pregnant and lactating women (currently breast-feeding or less than one year after delivery although not breast-feeding), women of childbearing potential who are not guaranteed effective contraception during the study, planning pregnancy or donating eggs or sperm within 6 months after the last dose.
* History of drug abuse or drug addicts.
* Subjects may not be able to complete the study duo to poor compliance or other reasons, or unsuitable for the study by the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 months
  overall remission rate, including complete remission without minimum residual disease (CRMRD-), complete remission (CR), complete remission with incomplete hematologic recovery (CRi), complete remission without platelet recovery (CRp), partial remission (PR).
composite complete remission (CRc) rate | up to 24 months.
  CRc rate is defined as the rate of all complete and incomplete remission (CRMRD-+CR+CRp+CRi).

SECONDARY OUTCOMES:
RFS | up to 24 months
  relapse-free survival, for patients achieving a complete remission, defined as the interval from the date of first documentation of a leukemia free state to date of recurrence, treatment failure, death due to any cause or last contact of the end-of-study follow up, which ever occurs first.
EFS | up to 24 months
  event-free survival, EFS is defined as the time from the date of enrollment until the date of documented relapse from CR, CRp or CRi, treatment failure, death from any cause or last contact of the end-of-study follow-up, whichever occurs first.
OS | up to 24 months
  overall survival, OS is defined as time from the date of enrollment until the date of death from any cause. For a subject who is not known to have died buy the end-of-study follow-up, OS is censored at the date of last contact.
duration of CR remission | up to 24 months
  DOR-CR is defined as the time from the date of first CR, CRp, CRi until the date of documented relapse.
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | up to 24 months
  safety and tolerability of investigational product assessed as the number of participants experience adverse events (AEs, CTCAE 5.0) or abnormalities in vital signs, laboratory tests, or electrocardiograms.
Cmax,ss | at the end of Cycle 1 (each cycle is 28 days)
  Peak plasma concentration at steady state
Cmin,ss | at the end of Cycle 1 (each cycle is 28 days)
  Minimum plasma concentration at steady state
Cav,ss | at the end of Cycle 1 (each cycle is 28 days)
  The average steady-state plasma concentration
AUCss | at the end of Cycle 1 (each cycle is 28 days)
  The area under the plasma concentration at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, MD. PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No